CLINICAL TRIAL: NCT07236580
Title: Is There Efficacy of Adding Buteyko Breathing to Approach of Smoking Hygiene on Dysfucntion of Eustachian Tube and Lung Functions in Adolescnets Who Are Passively Exposed to Tobacco Smoke?
Brief Title: Buteyko Breathing and Approach of Smoking Hygiene: Effects on Dysfucntion of Eustachian Tube and Lung Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-50
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Smoking; Eustachian Tube Dysfunction
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): in this group, we will include 20 adolescents who are usually exposed to tobacco smoke passively in house from smoking parent or household members. these adolescents will complain chronic dysfunction of their Eustachian Tube (chronic obstructive dysfucntion) . adolescents will receive smoking hyeigne approach for 6 months.This group will additionally receive Buteyko Breathing 30-minute apprach (this appraoch will be appleid by patients all days weekly, except fridays, for 6 months).
  Interventions: Behavioral: Buteyko breathing plus smoking hyeigne approach
- group number 2 (Active Comparator): in this group, we will include 20 adolescents who are usually exposed to tobacco smoke passively in house from smoking parent or household members. these adolescents will complain chronic dysfunction of their Eustachian Tube (chronic obstructive dysfucntion) . adolescents will receive smoking hyeigne approach for 6 months.
  Interventions: Behavioral: smoking hygiene appraoch

INTERVENTIONS:
Behavioral: Buteyko breathing plus smoking hyeigne approach — in this group, we will include 20 adolescents who are usually exposed to tobacco smoke passively in house from smoking parent or household members. these adolescents will complain chronic dysfunction of their Eustachian Tube (chronic obstructive dysfucntion) . adolescents will receive smoking hyeigne approach for 6 months.This group will additionally receive Buteyko Breathing 30-minute apprach (this appraoch will be appleid by patients all days weekly, except fridays, for 6 months).
  Arms: group number 1
Behavioral: smoking hygiene appraoch — in this group, we will include 20 adolescents who are usually exposed to tobacco smoke passively in house from smoking parent or household members. these adolescents will complain chronic dysfunction of their Eustachian Tube (chronic obstructive dysfucntion) . adolescents will receive smoking hyeigne approach for 6 months.
  Arms: group number 2

SUMMARY:
adolescents are usually exposed to tobacco smoke passively. this can reduce their lung functions and negatively impact functions of Eustachian tube. The solution is to lower rates to tobacco exposure and use the support of Buteyko Breathing

DETAILED DESCRIPTION:
in this study, we will randolmly recruit 40 adolescents who are usually exposed to tobacco smoke passively in house from smoking parent or household members. these adolescents will complain chronic dysfunction of their Eustachian Tube (chronic obstructive dysfucntion) . adolescents will be catagorized to one of both groupsl, group I or group II (N=20 patient in the group). Both groups will receive smokinh hyeigne approach for 6 months. Group I will additionally receive Buteyko Breathing 30-minute apprach (this appraoch will be appleid by patients all days, except fridays, weekly for 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Dysfucntion of Eustachian Tube (obstructive chronic form)
* adolescents with passive tobacco exposure from smoking parent or household member
* adolscent participants whose parents approve the participation

Exclusion Criteria:

* cardiac problem
* chest disease
* renal/hepatic disease

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Eustachian Tube dyafucntion questionaire | it will be measured after 6 months
  it is a questionaire contain 7 items

SECONDARY OUTCOMES:
percentage of change in type of tympanmetery | it will be measured after 6 months
  it will assess percenatge of type c tympanometry
forced vital capcity | it will be measured after 6 months
  it is a pulmaonry fucntion test
force expiratory volume (FEV1) | it will be measured after 6 months
  it will be mesured in the first second of expiration as a pulmaonry fucntion test
FEV1/FVC | it will be measured after 6 monthd
  it is a pulmaonry fucntion test
physical summary of parent form child health questinaire | it will be measured after 6 months
  it will assess quality of life
mental summary of parent form child health questinaire | it will be measured after 6 months
  it will assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt